CLINICAL TRIAL: NCT03705741
Title: The Efficacy of Light-to-moderate Resistance Training in Sedentary Pregnant Women: a Randomized Controlled Study
Brief Title: The Efficacy of Light-to-moderate Resistance Training in Sedentary Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 In summary, 48 persons were included.
Sponsor: Värmland County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Ylva Karolina Petrov Fieril, Principal Investigator, Fysiotherapist, PhD, Värmland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/246
Record Dates: First submitted 2018-10-03; First posted 2018-10-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy Related; Sedentary Lifestyle
Keywords: pregnancy; exercise; public health; randomized controlled trial
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Opaque sealed envelopes, which are randomly picked out before the meeting with each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Resistance exercise twice a week
  Interventions: Behavioral: Resistance exercise
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Resistance exercise — Resistance exercise twice a week during pregnancy week 23-34.
  Arms: Exercise group

SUMMARY:
Maintaining a physically active lifestyle is associated with many health benefits, including lower risk of cardiovascular disease, diabetes, hypertension, some type of cancer, and depression . Pregnant, healthy women are recommended to do 30 minutes or more of light to moderate exercise a day, although most women in the Western world do not follow current recommendations and decrease their exercise level.

Benefits of exercise during pregnancy are several, including a protective effect against the development of gestational diabetes mellitus, reduced pregnancy related low back pain, and risk of caesarean delivery. On the contrary, a recent review concludes that sedentary behaviors are associated with higher levels of C Reactive Protein and LDL Cholesterol, a larger newborn abdominal circumference, and macrosomia.

Previous studies show that exercise during pregnancy is associated with improvements in psychological well-being among previously sedentary women.

Only a few RCT's have studied resistance exercise during pregnancy. These studies have found reduced fatigue and reduced need of insulin among women with gestational diabetes mellitus who did resistance exercise, with no adverse effects on fetus or the pregnant woman.

The aim of this study is to evaluate the efficacy of regular light -to-moderate resistance exercise among sedentary pregnant woman, with regard to fatigue, health related quality of life, pain location and intensity, body weight gain, blood pressure, and childbirth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy and ≥18 of age
* Ability to understand verbal and written Swedish
* Inclusion during gestational week 20+0-20+6.

Exclusion Criteria:

* Follows the recommendation regarding contraindications according to the American Collage of Obstetricians and Gynecologists 2002
* Severe pain from the pelvic or the back
* Regular exercise >150 minutes per week the last six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | Register at gestational week 22 and 34
  Visual Analogue Scale (VAS) 0-100 millimeters. It is a psychometric scale and measure self-reported fatigue from 0, "no fatigue" to 100, "very great fatigue". The scale is a streight horizontal line.

SECONDARY OUTCOMES:
Change in anxiety / depression | Register at gestational week 22 and 34
  Visual Analogue Scale (VAS) 0-100 millimeters. It is a psychometric scale and measure self-reported anxiety/depression from 0, "no anxiety/depression" to 100, "very great anxiety/depression". The scale is a streight horizontal line.
Change in pain | Register at gestational week 22 and 34
  Visual Analogue Scale (VAS) 0-100 millimeters. It is a psychometric scale and measure the intensity of pain from 0, "none pain" to 100, "extreme amount of pain". The scale is a streight horizontal line.
Change in Health Related Quality of Life | Register at gestational week 22 and 34
  Visual Analogue Scale (EQ-VAS). Mark health status on the day on a 20 centimeters vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Change in blood pressure | From perinatal records. Registered at gestational week 22 and 34
  Systolic and Diastolic
Change in weight gain | from perinatal records. Registered at gestational week 22 and 34
  kilogram
Gestational Diabetes Mellitus (GDM) | from perinatal records. Registered at gestational week 34
  Development of GDM
Change in exercise | Registered at gestational week 22 and 34
  Minutes a day. (Walks, light, moderate, vigorous intensity).
Birth weight | from perinatal records at birth (gestational week 40)
  kilogram
Birth length | from perinatal records at birth (gestational week 40)
  centimeters
Gestational age | From perinatal records at birth (gestational week 40)
  days
Acute cesarean section | from perinatal records at birth (gestational week 40)
  rate
Macrosomia | from perinatal records at birth (gestational week 40)
  rate of birth with macrosomia

CONTACTS AND LOCATIONS:
Locations (1):
- Fysioterapimottagningen Gripen, Karlstad, Sweden

IPD SHARING:
Plan to Share IPD: No